CLINICAL TRIAL: NCT02619318
Title: Balancing Everyday Life - A Lifestyle Intervention for People With Psychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Mona Eklund, Professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEL (ViB)
Record Dates: First submitted 2015-11-20; First posted 2015-12-02 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Major Psychiatric Disorder
Keywords: Balancing Everyday Life (BEL); activity-based lifestyle intervention; standard occupational therapy

ARMS (2):
- The Balancing Everyday Life (BEL) intervention (Experimental): The BEL was developed on the basis of previous research on lifestyle interventions made by our own group and other researchers [1, 2]. It is a group-based programme (5-8 participants) with 12 sessions, one session a week, and 2 booster sessions with two-week intervals. The themes for the group sessions are, e.g., activity balance, healthy living, work-related activities, and social activities. Each session contains a main group activity and a home assignment to be completed between sessions. The main group activity starts with analysing the present situation and proceeds with identifying desired goals and finding strategies for how to reach them. The home assignment is aimed at testing one of the proposed strategies. Self-analysis, setting goals, finding strategies and evaluating the outcome of tested strategies form a process for each session, but also for the BEL intervention as a whole.
  Interventions: Behavioral: Balancing Everyday Life (BEL)
- Care as usual (standard occupational therapy) (Active Comparator): Standard occupational therapy involves support to open-market employment and support in managing everyday life in general.
  Interventions: Behavioral: Care as usual (generally standard occupational therapy)

INTERVENTIONS:
Behavioral: Balancing Everyday Life (BEL)
  Arms: The Balancing Everyday Life (BEL) intervention
Behavioral: Care as usual (generally standard occupational therapy)
  Arms: Care as usual (standard occupational therapy)

SUMMARY:
This is a RCT study, aiming at evaluating the effectiveness of the Everyday Life in Balance (BEL) intervention.

The intervention: The BEL was developed on the basis of previous research on lifestyle interventions made by the current research group and other researchers . It is a group-based programme (5-8 participants) with 12 sessions, one session a week, and 2 booster sessions with two-week intervals. The themes for the group sessions are, e.g., activity balance, healthy living, work-related activities, and social activities. Each session contains a main group activity and a home assignment to be completed between sessions. The main group activity starts with analysing the present situation and proceeds with identifying desired goals and finding strategies for how to reach them. The home assignment is aimed at testing one of the proposed strategies. Self-analysis, setting goals, finding strategies and evaluating the outcome of tested strategies form a process for each session, but also for the BEL intervention as a whole. After completed BEL, the participants will have developed an ability to reflect on their own situation and have strategies for changing their everyday life in a desired direction, such that they feel their everyday life has a satisfactory balance between rest and work, secluded and social activities, etc.

The BEL intervention is led by occupational therapists. They take part in a specifically developed two-day education and follow the BEL manual [7]. They also participate in a web-based discussion forum where they can seek support from the researchers and/ or other BEL occupational therapists.

Selection of units and participants: On the basis of blocks of four units, two are randomized to the BEL and two to the control condition, which is care as usual (CAU) and generally means standard occupational therapy. Occupational therapists in the units select participants based on the patients' needs for a lifestyle intervention and being likely to benefit from a group intervention. The same criteria are applied in the BEL units and the CAU units.

Power analysis: The investigators desire 120 participants from each group. This will also allow for analysis of subgroups.

Instruments: A number of self-report instruments tapping satisfaction with daily occupations, well-being, perceived worker role, social interaction, recovery etc., will be used, supplemented with qualitative interviews.

Procedure: As the intervention starts, the attendees answer questionnaires about their personal situation regarding. Subsequently, the BEL is implemented in the units randomised to that condition. After 16 weeks of intervention (including the booster sessions), the measurements are repeated. A follow-up is then made after another six months. The same data collection is made at corresponding time points in the comparison units.

Additional qualitative interviews are made in the intervention units, with strategically selected participants (attendees and staff) to get a deeper picture of the intervention process and its implications.

When the research project is finished, the comparison units will be given the opportunity to go through the intervention.

Analyses: The primary analysis concerns differences in outcomes between the BEL group and the CAU group. Analyses of the qualitative interviews, by means of grounded theory, will yield a more detailed description of the BEL and its implications, as perceived by both attendees and staff.

Current state of the study: The project is in the initial phase and the first units were recruited in late 2012. At present, 24 units have been randomized to either condition. The second measurements (after completed BEL) have just been completed and follow-ups will continue until mid-2016, as will qualitative interviews. Analysing data and reporting results will continue until late 2018.

By including 60 participants in each group the studies will be able to detect a medium effect size (ES=0.4), which would be a difference of clinical and practical significance.

Age, gender and being of foreign origin will be considered as covariates, along with other socioeconomic factors such as family situation, educational level and money at one's disposal. Other factors that should be considered are the participant's functional status and diagnoses. Research has not shown that diagnosis per se plays any substantial role in the outcome of psychiatric rehabilitation, for the course of a psychiatric disability or for how people perceive their everyday occupations, but this should be investigated further because the evidence is inconclusive. Level of functioning, level of psychopathology, and negative symptoms have indeed been shown to be of importance for outcomes of psychiatric rehabilitation. Therefore, this project will also control for factors related to diagnosis and functional status.

DETAILED DESCRIPTION:
Balancing Everyday Life - evaluation of the effectiveness of an activity-based lifestyle intervention for people with psychiatric disorders

This is a RCT study, evaluating the effectiveness of the Everyday Life in Balance (BEL) intervention.

The intervention: The BEL was developed on the basis of previous research on lifestyle interventions made by the current research group and other researchers. Other important sources of inspiration were descriptive studies on everyday life among people with severe mental illness. It is a group-based programme (5-8 participants) with 12 sessions, one session a week, and 2 booster sessions with two-week intervals. The themes for the group sessions are, e.g., activity balance, motivation, healthy living, work-related activities, leisure and social activities. Each session contains a brief educational section, a main group activity and a home assignment to be completed between sessions. The main group activity starts with analysing the present situation and proceeds with identifying desired goals and finding strategies for how to reach them. The home assignment is aimed at testing one of the proposed strategies. The next-coming session starts with looking back at the home assignment, and depending on the outcome, goals may need to be revised. Self-analysis, setting goals, finding strategies and evaluating the outcome of tested strategies form a process for each session, but also for the BEL intervention as a whole. After completed BEL, the participants will have developed an ability to reflect on their own situation and have strategies for changing their everyday life in a desired direction, such that they feel their everyday life has a satisfactory balance between rest and work, secluded and social activities, etc.

The BEL intervention is led by occupational therapists. They take part in a specifically developed two-day education and follow the BEL manual. They also participate in a web-based discussion forum where they can seek support from the researchers and/ or other BEL occupational therapists.

Selection of units and participants: Units in both county council-based psychiatry (outpatient units within general psychiatry and psychosis care) and community-based activity centers (CBACs) in four counties in south Sweden have been invited. Cluster randomization is used to assign the units to the BEL or the control condition. On the basis of blocks of four units, two are randomized to the BEL and two to the control condition, which is care as usual (CAU). CAU generally means standard occupational therapy. Four categories of participants will be recruited: a) BEL participants from county-council-based psychiatry; b) BEL participants from community-based psychiatry; c) CAU participants from county-council-based psychiatry; and d) CAU participants from community-based psychiatry. Occupational therapists in the units select participants based on the patients' needs for a lifestyle intervention and being likely to benefit from a group intervention. The same criteria are applied in the BEL units and the CAU units.

Power analysis: The investigators based the power calculation on the Satisfaction with Daily Occupations (SDO) scale. A previous study found a mean difference of 0.5 points on the SDO between groups of people with mental illness who had varying structure to their everyday life. Based on the means and standard deviations from that study, the analysis pointed to 41 participants in each condition as the desired sample size to detect a difference on the SDO of 0.5 with 80% power at p<0.05. The investigators still desire 60 participants from each group (a - d above) since no solid base for a power calculation exists in the field. In all 240 participants are thus sought, 60+60 receiving the BEL and 60-60 receiving CAU.

The following instruments are used:

Rosenberg's self-esteem scale: Positive and negative attitudes towards the self; Global Assessment of Functioning (GAF): Symptom severity and psychosocial functioning; Satisfaction with Daily Occupations and Balance (SDO-B): Satisfaction with everyday occupation and occupational balance; Occupational Value with pre-defined items (OVal-pd): Perceived value with daily occupation; Pearlin's Mastery Scale: Self-mastery; Medical Outcomes Short Form (SF-36) (1st item): Self-rated Health; Manchester Short Assessment of Quality of Life (MANSA): Quality of life; Interview Schedule for Social Interaction (ISSI): The social network; Worker Role Self-assessment (WRS): Attitudes and expectations concerning the worker role; "Making decisions": Empowerment; Client Satisfaction Questionnaire (CSQ): Satisfaction with the intervention; Estimating Perceived Meaning in Day Centers (EPM-DC): Characteristics of day centers; Questionnaire of Personal Recovery (QPR): Recovery from mental illness; Fidelity scale: Fidelity to the intervention.

In addition, consequences of the intervention will be reflected in qualitative interviews with users and staff. Another important part of the data collection will be to make a detailed description of the CAU provided in the comparison units.

Procedure: As the intervention starts, the attendees answer questionnaires about their personal situation regarding satisfaction with daily occupations, well-being, perceived worker role, social interaction, recovery etc. Subsequently, the BEL is implemented in the units randomised to that condition. After 16 weeks of intervention (including the booster sessions), the measurements are repeated. A follow-up is then made after another six months. The same data collection is made at corresponding time points in the comparison units.

Additional qualitative interviews are made in the intervention units, with strategically selected participants (attendees and staff) to get a deeper picture of the intervention process and its implications.

When the research project is finished, the comparison units will be given the opportunity to go through the intervention.

Analyses: The primary analysis concerns differences in outcomes between the intervention and the control group (a+b versus c+d above), at the unit level (characteristics of the CBACs) and the individual level (perceptions of worker role, satisfaction, well-being etc.), and the stability of such outcomes. The sample size will also allow for comparison between community-based and county-council-based BEL. Since measuring characteristics of CBACs is not of relevance for county council-based psychiatry, the comparison at the unit level will only concern community-based psychiatry.

Analyses of the qualitative interviews, by means of grounded theory [10], will yield a more detailed description of the BEL and its implications, as perceived by both attendees and staff.

Current state of the study: The project is in the initial phase and the first units were recruited in late 2012. At present, 24 units have been randomized to either condition. The second measurements (after completed BEL) have just been completed and follow-ups will continue until mid-2016, as will qualitative interviews. Analysing data and reporting results will continue until late 2018.

Methodological considerations By including 60 participants in each group the studies will be able to detect a medium effect size (ES=0.4), which would be a difference of clinical and practical significance.

Self-rating instruments are used and it is important to consider whether these produce reliable data when used with people with SMI, particularly since many in the target group have cognitive problems. However, research has shown that self-ratings of psychological factors were valid and reliable among people with schizophrenia, also those with a poor insight into their mental illness.

Age, gender and being of foreign origin will be considered as covariates, along with other socioeconomic factors such as family situation, educational level and money at one's disposal. Other factors that should be considered are the participant's functional status and diagnoses. Research has not shown that diagnosis per se plays any substantial role in the outcome of psychiatric rehabilitation, for the course of a psychiatric disability or for how people perceive their everyday occupations, but this should be investigated further because the evidence is inconclusive. Level of functioning, level of psychopathology, and negative symptoms have indeed been shown to be of importance for outcomes of psychiatric rehabilitation. Therefore, this project will also control for factors related to diagnosis and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Having a major psychiatric disorder,
* age of 18-65 years,
* in need of a lifestyle intervention (as assessed by an occupational therapist)

Exclusion Criteria:

* Comorbidity of dementia or developmental disability,
* substance use disorder as main diagnosis, acute psychosis,
* not being able to communicate in Swedish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in occupational satisfaction and balance as measured by the Satisfaction with Daily Occupations and Balance (SDO-B) scale | Change from baseline to completed intervention, an average of 16 weeks
  Perceived balance between one's everyday activities
Change in valued activities as measured by the Occupational Value with pre-defined items ( OVal-pd) | Change from baseline to completed intervention, an average of 16 weeks
Change in personal recovery as measured by the Questionnaire of Personal Recovery (QPR) | Change from baseline to completed intervention, an average of 16 weeks
  Personal perceptions of recovery, although clinical recovery has not been accomplished

SECONDARY OUTCOMES:
Change in quality of life as measured by the Manchester Short Assessment of Quality of Life (MANSA) | Change from baseline to completed intervention, an average of 16 weeks
Change in self-mastery as measured by Pearlin's Mastery Scale | Change from baseline to completed intervention, an average of 16 weeks
  Sense of being able to influence one's life situation
Change in self-esteem as measured by Rosenberg's Self-esteem Scale | Change from baseline to completed intervention, an average of 16 weeks

OTHER OUTCOMES:
Satisfaction with the intervention received, as measured by the Client Satisfaction Questionnaire (CSQ) after the 16-week intervention | At completion of the 16-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mona Eklund, PhD, prof., Principal Investigator — Lund University
Locations (1):
- Skåne Psychiatry, Lund, Skåne County, Sweden

REFERENCES:
- [Derived] Argentzell E, Backstrom M, Lund K, Eklund M. Exploring mediators of the recovery process over time among mental health service users, using a mixed model regression analysis based on cluster RCT data. BMC Psychiatry. 2020 Oct 30;20(1):520. doi: 10.1186/s12888-020-02924-2. PMID 33126873
- [Derived] Hultqvist J, Lund K, Argentzell E, Eklund M. Predictors of clinically important improvements in occupational and quality of life outcomes among mental health service users after completion and follow-up of a lifestyle intervention: multiple regression modelling based on longitudinal data. BMC Psychol. 2019 Dec 17;7(1):83. doi: 10.1186/s40359-019-0359-z. PMID 31847910
- [Derived] Eklund M, Tjornstrand C, Sandlund M, Argentzell E. Effectiveness of Balancing Everyday Life (BEL) versus standard occupational therapy for activity engagement and functioning among people with mental illness - a cluster RCT study. BMC Psychiatry. 2017 Nov 9;17(1):363. doi: 10.1186/s12888-017-1524-7. PMID 29121882